CLINICAL TRIAL: NCT01083264
Title: Open-label, Randomized, Crossover Study to Investigate the Relative Bioavailability of Transdermally Administered Ethinylestradiol (EE) and Gestodene (GSD) After Repeated Applications of a Fertility Control Patch Containing 0.55 mg Ethinylestradiol and 2.1 mg Gestodene to 3 Different Application Sites (Buttocks, Arm Versus Abdomen) in Healthy Young Female Subjects
Brief Title: Relative Bioavailability, Transdermally Administered EE and GSD, 3 Applications Sites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 91608; 2009-011151-52 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Contraception
Keywords: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)
- Arm 2 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)
- Arm 3 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)

INTERVENTIONS:
Drug: Gestodene/EE Patch (BAY86-5016) — Transdermal Patch, 0.55mg Ethinylestradiol + 2.1mg Gestodene, 4x7 days patch wearing period, patch-free interval of 7 days, application site: buttocks
  Arms: Arm 1
Drug: Gestodene/EE Patch (BAY86-5016) — Transdermal Patch, 0.55mg Ethinylestradiol + 2.1mg Gestodene, 4x7 days patch wearing period, patch-free interval of 7 days, application site: arm
  Arms: Arm 2
Drug: Gestodene/EE Patch (BAY86-5016) — Transdermal Patch, 0.55mg Ethinylestradiol + 2.1mg Gestodene, 4x7 days patch wearing period, patch-free interval of 7 days, application site: abdomen
  Arms: Arm 3

SUMMARY:
Influence of different application sites on the blood levels after administration of a fertility control patch

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* Age 18-45 years
* Body mass index (BMI) 18-30kg/m²
* At least 3 months since delivery, abortion, or lactation before the first screening examination
* Ability to understand and follow study-related instructions
* Willingness to accept the synchronizing cycle and to use non-hormonal methods of contraception after starting the synchronizing cycle and during the treatment periods

Exclusion Criteria:

* Contra-indications for use of combined (estrogen/progestin) contraceptives (e.g. history of venous/arterial disease, liver disorders, migraine)
* Skin diseases with suspected alteration of dermal resorption and /or increased risk for dermal intolerance
* Regular use of medicines other than contraceptives
* Smokers (at the age of 31 to 45 years)
* Clinically relevant findings (e.g. blood pressure, physical and gynecological examination, laboratory examination)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
AUC(0-168) for EE and Gestodene during week 4 of each treatment period | Week 4 of each treatment period ( 3 periods)

SECONDARY OUTCOMES:
Pharmacokinetic parameters of EE and GSD: Cmax, Cmin, Cav, tmax, t1/2 obtained during week 4, Ctrough obtained at the end of each week | Week 1-5 of each treatment period
Adverse Events | Week 1-5 of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany